CLINICAL TRIAL: NCT06696599
Title: Serum and Corporal Irisin Level and Its Correlation With Erectile Function in Diabetic Obese Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Islam Mohamed Abdelrahman fahem, Resident doctor, Assiut University
Other Study IDs: Irisin in erectile dysfunction
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Serum and Corporal Irisin in Diabetic Patients With Erectile Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Serum and corporal irisin in diabetic patients: Penil duplex ,serum irisin ,corporal irisin
  Interventions: Procedure: Serum and corporal irisin
- Serum irisin in normal persons: Serum irisin

INTERVENTIONS:
Procedure: Serum and corporal irisin — measure serum and corporal irisin
  Groups: Serum and corporal irisin in diabetic patients

SUMMARY:
Obese and diabetic men constitute a huge fraction of ED patients. There is established relation between both obesity ,diabetes and ED through multiple neuroendocrine and vascular players .

A limited number of serum biomarkers are available for ED with diabetic patients. These are biomarkers often used for endothelial dysfunction, inflammation and oxidative stress. Serum E-selectin, endothelial progenitor cell (EPC), endothelial micro particle (EMP), tumour necrosis factor / interleukin-10 (TNF-a / IL-10), nitric oxide (NO), MDA (malondialdehyde) and lipoprotein (a) are the most used biomarkers in this population.

DETAILED DESCRIPTION:
Obese and diabetic men constitute a huge fraction of ED patients. There is established relation between both obesity ,diabetes and ED through multiple neuroendocrine and vascular players .

A limited number of serum biomarkers are available for ED with diabetic patients. These are biomarkers often used for endothelial dysfunction, inflammation and oxidative stress. Serum E-selectin, endothelial progenitor cell (EPC), endothelial micro particle (EMP), tumour necrosis factor / interleukin-10 (TNF-a / IL-10), nitric oxide (NO), MDA (malondialdehyde) and lipoprotein (a) are the most used biomarkers in this population.

Irisin is a novel skeletal muscle- and adipose tissue-secreted peptide. It is conventionally regarded as an adipomyokine and is a cleaved fragment of Fibronectin type III domain containing protein 5 (FNDC5). It is involved in the browning of white adipose tissue, glucose tolerance, and reversing of metabolic disruptions.

Irisin exerts a direct vascular protective effect on endothelial function:- The mechanism for this protective effect of irisin appeared to be related AMP activated protein kinase and endothelial NO synthase (AMPK-eNOS) signaling pathway activation.Irisin enhanced NO production and phosphorylation of AMPK, Akt, and eNOS in endothelial cells.

According to a recently published study, The use of exogenous irisin is thought to alleviate endothelial dysfunction in T2DM by reducing oxidative / nitrative stresses. Therefore, it can be used in the future to eliminate the vascular complications of diabetes.Although the relationship between T2DM, endothelial dysfunction and irisin has been demonstrated in many previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Age of patients 30-50 years old .
* patients with type ll diabetes mellitus .
* patients on oral hypoglycemic medications .
* Non responders PDEI-5 ED patients

Exclusion Criteria:

* Age of patients above 60 years old .
* patients with type l diabetes mellitus on insulin .
* patients with hypogonadism .

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Cross sectional
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Association between irisin and erectile function in 50 patients 40 patients complaint from erectile dysfunction and 10 patients have good erection | 2 years
  Measurement serum and corporal irisin in diabetic patients with erectile dysfunction

IPD SHARING:
Plan to Share IPD: Undecided